CLINICAL TRIAL: NCT04919031
Title: Inspiratory Muscle Trainer Impact on Post Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) COVID-19 Hypertensive Patients With Long Term Persistent Symptoms
Brief Title: Inspiratory Muscle Trainer and Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) COVID-19 Persistent Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ebtesam Nabil, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/003228
Record Dates: First submitted 2021-06-07; First posted 2021-06-09 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Covid19; Hypertension; Corona Persistent Symptoms
MeSH Terms: conditions — COVID-19; Hypertension

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study (Experimental): Inspiratory muscle trainer plus diaphragmatic release and traditional medications
  Interventions: Device: Inspiratory muscle trainer; Other: diaphragmatic release
- control (Active Comparator): inspiratory muscle trainer plus traditional medications
  Interventions: Device: Inspiratory muscle trainer

INTERVENTIONS:
Device: Inspiratory muscle trainer — POWER breathe IMT is a drug-free, hand-held breathing training device. The medical term for this type of breathing training is Inspiratory Muscle Training, or IMT. POWER breathe IMT exercises the main muscles you use to breathe in, primarily your diaphragm and intercostal
Other: diaphragmatic release — diaphragmatic release is a manual technique use for restoring the ability of the diaphragm to go through a full range of motion
  Arms: study

SUMMARY:
Inspiratory muscle training considered as safe and valid method to improve respiratory muscle strength and functional capacity among uncountable conditions which could improve post COVID-19 persistent symptoms including but not limited to respiratory muscle strength, diminishing dyspnea, enhance blood oxygenation, and patient's functional capacity and quality of life.

DETAILED DESCRIPTION:
The current COVID-19 pandemic will place enormous pressure on healthcare systems around the world. The COVID-19 pandemic continues to dominate our daily lives with large numbers of people are predicted to become critically ill with acute respiratory distress syndrome and will require management in intensive care units. Unfortunately, it is expected that COVID-19 will persist as a major challenge for the delivery of medical care for a long while to go. High levels of physical, cognitive, and psychosocial impairments can be anticipated and persist after discharging from hospitals. Growing data shows a higher risk of COVID-19 infections and complications in people with high blood pressure affecting between 30% to 50% of the patients.

Intensive care unit- acquired weakness is very common after ARDS (COVID 19) which confers a major determinant of poor long-term functional, respiratory and psychological outcome.

Patients with coronavirus disease (COVID-19) are described as exhibiting oxygen levels incompatible with life with dyspnea. Pulse oximeter is valid device used to assess oxygen level in the blood as well as the pulse rate. As case numbers grow, neurological symptoms have been reported with increasing the frequency of corona virus infection, including those of autonomic dysfunction. It was reported that many patients developed postural tachycardia syndrome (POTS) several months after confirmed SARSCoV- 2 infection especially those with cardiovascular risk factors. Based on knowledge from the multiple systemic complications associated with Covid-19, it is reasonable to suggest that most patients, especially those who underwent prolonged hospitalization with one or more cardiovascular risk factor, will need a multi professional rehabilitation program.

Respiratory rehabilitation aims to improve quality of life by managing dyspnea, improving exercise tolerance and increasing functional capacity. After initial recovery from Covid-19, especially for those who required hospitalization in ICU, it is possible that some patients may experience respiratory muscle dysfunction, as well as pulmonary restriction or obstruction to varying extents, affecting peripheral muscle function and respiratory conditioning.

Several previous studies explained that inspiratory muscle training (IMT) is a feasible and safe modality in patients with respiratory muscle dysfunction which approve its efficacy in enhancing respiratory muscle strength, improving aerobic capacity, and diminishing dyspnea among patients suffering from COVID 19.

ELIGIBILITY:
Inclusion Criteria:

* sixty non hospitalized negative post covid-19
* men
* cigarette smokers
* 40-60 years old
* stage II Hypertensive (160-179 / 100-109 mmHg)
* Oxygen saturation less than 94%
* Severity of disease (Moderate Covid-19 affection)
* Body mass index (BMI) ranged from 25 to 29.9 kg/m2
* hemodynamically stable
* at least 4 weeks since first COVID-19 swab at time of screening

Exclusion Criteria:

* Patients with red flag indicators as chest pain, critical drop of oxygen saturation which require oxygen supply, severe level of hypoxia (blue lips)
* Unconscious patient
* Positive covid-19 patients
* Patients with cognitive impairment
* End-stage of chronic diseases
* BMI more than 30 kg/m2
* History of other cardiovascular disease as coronary artery disease, valvular heart disease, cardiac arrhythmias, congestive heart failure, myocardial infarction, stroke, transient ischemic attack, or peripheral vascular disease
* Neurological, neuromuscular, and musculoskeletal limitations
* Current active infection
* Developmental disability or cognitive impairment that in the opinion of the investigator would preclude adequate comprehension of the informed consent form and/or ability to record the necessary study measurements.
* Participation in a clinical study or other type of research in the past 30 days

Ages: 40 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-11-23 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
maximal inspiratory pressure | 6 weeks
  For determining MIP, patients breathe through a flanged mouthpiece with nose clips in place. They are instructed to exhale to RV. At RV, a valve or shutter is closed, and the patient is coached to inhale as forcefully as possible. Maximum pull should be maintained for 1-2 seconds.

SECONDARY OUTCOMES:
sleeping quality scale | 6 weeks
  Consisting of 28 items, the SQS evaluates six domains of sleep quality: daytime symptoms, restoration after sleep, problems initiating and maintaining sleep, difficulty waking, and sleep satisfaction. Using a four-point, respondents indicate how frequently they exhibit certain sleep behaviors (0 = "few," 1 = "sometimes," 2 = "often," and 3 = "almost always").
  Scores on items belong to factors 2 and 5 (restoration after sleep and satisfaction with sleep) and are reversed before being tallied. Total scores can range from 0 to 84, with higher scores demoting more acute sleep problems.
Timed stair climbing | 6 weeks
  Total time to ascend and descend steps is recorded to the nearest 100th of a second. Lower values = better performance
6 minute walk test | 6 weeks
  The 6 Minute Walk Test is a sub-maximal exercise test used to assess aerobic capacity and endurance. The distance covered over a time of 6 minutes by meter is used as the outcome by which to compare changes in performance capacity.
modified medical research council (mMRC) scale (0-4) | 6 weeks
  The mMRC scale is a self-rating tool to measure the degree of disability that breathlessness poses on day-to-day activities on a scale from 0 to 4: 0, no breathlessness except on strenuous exercise; 1, shortness of breath when hurrying on the level or walking up a slight hill; 2, walks slower than people of same age on the level because of breathlessness or has to stop to catch breath when walking at their own pace on the level; 3, stops for breath after walking ∼100 m or after few minutes on the level; and 4, too breathless to leave the house, or breathless when dressing or undressing
Oxygen saturation | 6 weeks
  pulse ox meter used to assess peripheral oxygen saturation
dyspnea borg scale | 6 weeks
  This is a scale that asks you to rate the difficulty of your breathing. It starts at number 0 where your breathing is causing you no difficulty at all and progresses through to number 10 where your breathing difficulty is maximal
postural tachycardia syndrome | 6 weeks
  the heart rate measured by pulse oxy-meter which applied on the index finger
blood pressure (mmHg) | 6 weeks
  a sphygmomanometer will be used to measure the blood pressure (systolic and diastolic values)
lactate level | 6 weeks
  venous blood sample will be drawn to assess blood lactate level. normal blood lactate level equal or less than 1 mmol/l
fatigue severity scale (0-63) | 6 weeks
  The Fatigue Severity Scale (FSS) is a method of evaluating the impact of fatigue on patients. The FSS is a short questionnaire that requires the patient to rate his level of fatigue.
  The FSS questionnaire contains nine statements that rate the severity of the fatigue symptoms from 1 to 7, based on how accurately it reflects patient condition during the past week and the extent to which agree or disagree that statement
  * A low value (e.g., 1) indicates strong disagreement with the statement, whereas a high value (e.g., 7) indicates strong agreement.
  * A total score of less than 36 suggests suffering from fatigue. A total score of 36 or more suggests needing further evaluation by a physician
Patient health questionnaire (PHQ-9) | 6 weeks
  it is a reliable and valid measure of depression severity as it is a self reporting questionnaire from 1to 27. A low value (e.g.,1) indicates minimal depression while a high value (e.g., 27) indicates severe depression

CONTACTS AND LOCATIONS:
Overall Officials: Ebtesam N Nagy, doctoral, Principal Investigator — Cairo University
Locations (1):
- Faculty of Physical Therapy, Giza, Dokki, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: one year after study actual completion date